CLINICAL TRIAL: NCT01563094
Title: Bone Accrual and Hormones in Response to Lactation
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Principal Investigator, Sue Brown, Assistant Professor of Medicine, University of Virginia
Other Study IDs: 12441
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Lactation
Keywords: Bone Density; Lactation; Bone Turnover Markers
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective observational trial of healthy postpartum women to investigate changes in bone density and markers of bone turnover during lactation. The study hypothesis is that women who breast-feed 5 months or more will lose bone density and subsequently regain the bone density after weaning. This study seeks to define determinants of the regain in bone density.

DETAILED DESCRIPTION:
This is a prospective observational trial enrolling healthy postpartum women, ages 20 years and older with the intent to breast-feed from the UNC outpatient obstetrical clinics and the UVA outpatient obstetrical clinics. These women were studied at 3-5 visits in the year following their delivery to assess bone density, nutritional intake, exercise, and breast-feeding choices. The number of study visits depended on the timing of return of menses and interest in participating in the follow-up study (timepoints are: immediate postpartum, 3 months postpartum, return of menses, 6 months after return of menses and follow-up visit 6 months after final visit). Blood was taken for analysis of bone-related hormones, bone turnover and calcium homeostasis markers. The study focuses on women with extended lactation (at least 5 months of lactation) whereas women who cease lactation prior to 3 months will be the primary comparison group.

ELIGIBILITY:
Inclusion Criteria:

* age >20 at the time of delivery
* singleton pregnancy and
* <2 prior pregnancies that were >20 weeks gestation.

Exclusion criteria:

* maternal rheumatologic disorders
* maternal anorexia nervosa
* maternal endocrinologic disorders,
* medications known to affect bone density such as corticosteroids, thyroid hormone use, anticonvulsant therapy, bisphosphonates, long-term GnRH agonists use and calcitonin.
* Subsequent pregnancy during the study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postpartum women from outpatient obstetrical/gynecology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2003-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The association of change in bone density and change in IGF-1 axis hormones during lactation and weaning | ~Two Years

SECONDARY OUTCOMES:
The association of changes in bone density and change in bone turnover markers during lactation and weaning. | ~Two years

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — UVA
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD may be available by direct request of Principal Investigator.